CLINICAL TRIAL: NCT05859594
Title: The Effect of Laughter Yoga on Vasomotor Symptoms and Sleep Quality in Menopausal Women
Brief Title: The Effect of Laughter Yoga on Vasomotor Symptoms and Sleep Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Ahu AKSOY, Research Assistant, PhD, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 246
Record Dates: First submitted 2023-05-05; First posted 2023-05-16 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Vasomotor; Syndrome; Sleep
Keywords: vasomotor symptoms; sleep quality; menopause; laughter yoga; laughter therapy
MeSH Terms: conditions — Syndrome; Sleep Initiation and Maintenance Disorders | interventions — Laughter Therapy

STUDY DESIGN:
Intervention Model Description: Prospective, parallel, two arm, randomized controlled clinical trial
Who Masked: Outcomes Assessor
Masking Description: Statistical analysis of the data will be done by an expert independent of the research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (laughter yoga) group (Experimental): The intervention group will receive eight online laughter yoga sessions, two sessions per week for four weeks. In this study, the number of laughter yoga sessions was determined in line with the studies in the literature. Each laughter yoga session is planned to last approximately 40-45 minutes. Each session of laughter yoga consists of clapping and warm-up exercises, deep breathing exercises, childlike play and laughter.
  Interventions: Other: Laughter yoga
- Control group (No Intervention): The control group will receive no intervention for 4 weeks.

INTERVENTIONS:
Other: Laughter yoga — Although the history of laughter yoga dates back to ancient times, its use in medicine has become widespread in the 21st century, while it is used to reduce pain, anxiety, stress, depression and fatigue, it is also a method that can be used to accelerate immunity, quality of life, happiness, sleep quality and recovery.
  Other Names: Laughter therapy
  Arms: Experimental (laughter yoga) group

SUMMARY:
The research was planned as a prospective, randomized controlled experimental study to determine the effect of online laughter yoga applied to menopausal women on vasomotor symptoms (VMS) and sleep quality. Research Hypotheses ar below; H0: Online laughter yoga has no effect on VMS. H1: Online laughter yoga has an effect on VMS. H0: Online laughter yoga has no effect on sleep quality. H1: Online laughter yoga has an effect on sleep quality.

DETAILED DESCRIPTION:
The sample will consist of 82 menopausal women aged 40-60 years and experiencing at least one of the VMS. Intervention group: Online laughter yoga will be applied to women by a researcher who has an internationally approved certificate. The intervention group will receive eight online laughter yoga sessions, two sessions per week for four weeks. In this study, the number of laughter yoga sessions was determined in line with the studies in the literature. Each laughter yoga session is planned to last approximately 40-45 minutes. Each session of laughter yoga consists of clapping and warm-up exercises, deep breathing exercises, childlike play and laughter.

No intervention will be applied to the control group.

ELIGIBILITY:
Inclusion Criteria:

* - enrolled in the Menopause School,
* Signing the Informed Consent Form,
* Willing to participate in the research,
* Able to read and write Turkish,
* Open to communication,
* Those who are between the ages of 40-60 and have not experienced menstruation for at least one year,
* Experiencing at least one of the vasomotor symptoms
* A VMS severity of at least 4 according to the Visual Analog Scale,
* Not using drugs for the treatment of vasomotor symptoms,
* No chronic disease
* Regular laughter yoga is not practiced,
* Those who have not entered the menopause surgically,
* Women without psychiatric problems

Exclusion Criteria:

* - Not enrolled in Menopause School,
* Not signing the Informed Consent Form,
* Not willing to participate in the research,
* Cannot read and write Turkish,
* Unable to communicate
* Less than 40 years old, over 60 years old, experienced menstruation for at least one year,
* Not experiencing vasomotor symptoms,
* VMS severity is less than 4 according to the Visual Analog Scale,
* Using drugs for the treatment of vasomotor symptoms,
* Having a chronic disease,
* Regular laughter yoga practice
* Those who have surgically entered the menopause,
* Women with psychiatric problems

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 36 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scala (VAS) | change from baseline, at the end of 4th week of intervention.
  The Visual Analog Scale is used to measure the pain perceived by the person. There is a 10 cm mark on the one end of the scale, where there is no pain (zero), and on the other end there is the most severe (10) pain. Between the (100 mm.) part, the individual can indicate his or her pain by drawing a line, putting a dot or pointing. The distance from the point where there is no pain to the point marked by the individual is measured in centimeters, and the value found indicates the severity of the individual's pain. In this study, VAS will be used for hot flashes, night sweats and sweating experienced by women. Women will indicate where their situation is appropriate on this line by drawing a line or by placing a dot/mark.

SECONDARY OUTCOMES:
Sleep quality | change from baseline, at the end of 4th week of intervention.
  The Pittsburgh Sleep Quality Index (PUKI) will be used to assess sleep quality. PUKI sleep quality; subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleeping pills, and daytime dysfunction. Those with a total score above five on the PUKI are considered "poor", and those with a score of five or below are considered "good".

CONTACTS AND LOCATIONS:
Overall Officials: Ahu Aksoy Can, PhD, Principal Investigator — Mersin University Nursing Faculty
Locations (1):
- Mersin University, Yenişehir, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The effect of online laughter therapy on depression, anxiety, stress, and loneliness among nursing students during the Covid-19 pandemic — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC9477613/pdf/main.pdf